CLINICAL TRIAL: NCT06140862
Title: Ipsilateral Calf Muscle Weakness Induces Contralateral Radiculopathy , Where is the Clinical Biomechanics? "Part I"
Brief Title: Ankle Spine Syndrome "RAFFET Syndrome II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Noha Khaled Shoukry (Other)
Responsible Party: Sponsor-Investigator, Noha Khaled Shoukry, lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CUniv
Record Dates: First submitted 2023-11-15; First posted 2023-11-20 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Chronic Ankle Injuries; Chronic Low-back Pain; Lumbar Disc Herniation; Calf Muscle Weakness
Keywords: Ankle Spine Syndrome; Raffet Syndrome II; Contralateral Lumber Radiculopathy
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calf muscle exercise (Experimental): the initial treatment plane was open and closed chain strengthening exercises for the calf muscle. The strengthening exercises include; double leg calf raise (i.e., straight and bent knees), single leg calf raise (i.e., straight and bent knee), seated calf raise, and wall sit calf raise. Calf stretching exercises were added to maintain the flexibility of the muscle and its Achilles tendon. Gait training protocol was also performed for correction of chronically adapted abnormal gait pattern especially at the mid stance and terminal stance sub-phases of GC
  Interventions: Other: calf muscle strengthening and streching
- lower back exercise (Other): lumbar stabilization exercises, core strength training, myofascial release therapy for lower back, and stretching exercises for hamstring muscle.
  Interventions: Other: calf muscle strengthening and streching

INTERVENTIONS:
Other: calf muscle strengthening and streching — lumbar stabilization exercises, core strength training, myofascial release therapy for lower back, and stretching exercises for hamstring muscle.
  Other Names: lower back rehabilitation program

SUMMARY:
A case series aimed to describe a new clinical condition for the first time in the medical literature called Ankle Spine Syndrome or "RAFFET Syndrome II". This syndrome was reported in 6 patients (2 males and 4 females) out of 1000 patients with a history of chronic ankle injuries affecting their calf muscles' strength throughout the last 3 years. The patients suffered from unresolved CLBP with radiculopathy contralateral to their calf muscle atrophy (i.e., an ipsilateral calf muscle weakness induces contralateral lumbar radiculopathy) that did not respond to physical therapy or any medication for long.

DETAILED DESCRIPTION:
There is a large body of research performed to investigate the etiology of contralateral radiculopathy. However, limited information exists to determine its incidence, underlying pathomechanics, and strategies for management. Therefore, this case series aimed to describe a new clinical condition for the first time in the medical literature called Ankle Spine Syndrome or "RAFFET Syndrome II". This syndrome was reported in 6 patients (2 males and 4 females) out of 1000 patients with a history of chronic ankle injuries affecting their calf muscles' strength throughout the last 3 years. The patients suffered from unresolved CLBP with radiculopathy contralateral to their calf muscle atrophy (i.e., an ipsilateral calf muscle weakness induces contralateral lumbar radiculopathy) that did not respond to physical therapy or any medication for long. Open and closed chain strengthening exercises for the calf muscle were performed. The strengthening exercises include; double leg calf raise (i.e., straight and bent knees), single leg calf raise (i.e., straight and bent knee), seated calf raise, and wall sit calf raise. The patients' long-term back pain and function resolved greatly. By including lumbar stabilization exercises, core training, and myofascial release therapy, the symptoms resolved completely. Furthermore, with a follow-up after 6 months of a tailored home exercise program, the clinical outcome measures still resolved completely.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation of lumbar radicular pain (i.e., contralateral radiculopathy) was sharp, distinctive, shooting, or lancinating. It felt like a narrow band of pain (i.e., not more than 5-8 cm wide) throughout the length of the lower limb. It was experienced superficially and deeply.

They had back pain intensity scores that ranged from 8 to 10 indicating a severe degree of pain during dynamic activity while almost all patients scored zero while resting Our patients with this syndrome had functional disability scores that ranged from 10 to 22 indicating mild and moderate degrees of disability.

had a history of physical therapy visits for back pain and sciatica at many specialized centers

Exclusion Criteria:

* pain score less than 8 functional disability scores less than 10 red flags as tumor or osteoprosis or bone infection previous back surgery

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) known as Oswestry Low Back Pain Disability Questionnaire | six month
  It is a 10-section, self-report questionnaire to evaluate the impact of back pain on functional activities. Our patients in this syndrome had functional disability scores that ranged from 10 to 22 indicating mild and moderate degrees of disability. It is a valid, reliable and responsive clinical tool used to determine the level of functional disability associated with CLBP

SECONDARY OUTCOMES:
back pain was assessed using Numerical Pain Rating Scale (NPRS) | 6 month
  It is 11-point numeric scale ranges from zero that indicates "no pain" to 10 that indicates "the worst pain possible". The patients were asked to select a value that is most in line with the intensity of pain that they have experienced in the last 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Cairo University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided